CLINICAL TRIAL: NCT05356832
Title: Investigation of the Relationship Between Pelvic Floor Awareness and Urinary Incontinence in Young Athletes
Brief Title: Investigation of the Relationship Between Pelvic Floor Awareness and Urinary Incontinence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pinar Yasar (Other)
Responsible Party: Sponsor-Investigator, Pinar Yasar, Research assistant, Physiotherapist, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Other Study IDs: E 87432956-050.99-184902
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Pelvic Floor; Urinary Incontinence; Young Athletes
Keywords: pelvic floor; awareness; knowledge; urinary incontinence; athletes
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- continent: able to hold urine during sports
  Interventions: Diagnostic Test: Pelvic Floor Health Knowledge Quiz
- incontinent: leaking urine during sports
  Interventions: Diagnostic Test: Pelvic Floor Health Knowledge Quiz

INTERVENTIONS:
Diagnostic Test: Pelvic Floor Health Knowledge Quiz — It is a questionnaire to measure the knowledge level of the participants about pelvic floor health.
  Other Names: International Physical Activity Questionnaire-Short Form; International Consultation on Incontinence Questionnaire-Short Form; Incontinence Impact Questionnaire-7

SUMMARY:
There is no study in the literature examining the knowledge level and urinary symptoms of active athletes about the pelvic floor. The aim of this study is to determine the relationship between PTC awareness and incontinence in young athletes who engage in long-term and high-intensity activities that increase the risk of SUI.

ELIGIBILITY:
Inclusion Criteria:

18-25 years old Young athletes

Exclusion Criteria:

Having a neurological disorders

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young athletes studying at Süleyman Demirel University, Faculty of Sport Sciences
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire- Short Form | baseline
  The physical activity level is determined by recording the light, moderate and vigorous activities and sitting time of the person in the last 1 week.
Pelvic Floor Health Knowledge Quiz | baseline
  It is a questionnaire to measure the knowledge level of the participants about pelvic floor health.
International Urinary Incontinence Consultation Questionnaire-Short Form (ICIQ-SF) | baseline
  It is a questionnaire containing six questions to find out the frequency of urinary incontinence, during which activities it occurs, and how much the person is affected by this condition.
Incontinence Impact Questionnaire-7 | baseline
  It is a questionnaire consisting of 7 questions used in the evaluation of daily life effects due to incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Pinar YASAR, Study Director — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)